CLINICAL TRIAL: NCT06104995
Title: Effects of a Short Educational Video on Back Beliefs Among the General Population
Brief Title: Back Beliefs Among the General Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bern University of Applied Sciences (Other)
Collaborators: Haute Ecole de Santé Vaud (Other)
Responsible Party: Principal Investigator, Stefan Schmid, Deputy Head of Research at the Division of Physiotherapy and Head of Spinal Movement Biomechanics Group, Bern University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: BernUASBackBeliefs
Record Dates: First submitted 2023-10-16; First posted 2023-10-27 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Low Back Pain
Keywords: nonspecific low back pain; back beliefs; education
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will fill out online questionnaires. No outcome assessor will be present or in contact with the participants. The investigator that will analyse the data will not be aware of which participants are in which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Educational video on back beliefs (Experimental): Participants receive an educational video on back beliefs and its contributing factors.
  Interventions: Other: Interventional video
- Control Video Education (Experimental): Participants receive a neutral video about the back (e.g. anatomy of the back).
  Interventions: Other: Control video

INTERVENTIONS:
Other: Interventional video — The educational video comprises of health care professionals explaining the durability of the back against the popular belief that the back is fragile and the multifactorial nature of back pain.
  Arms: Interventional Educational video on back beliefs
Other: Control video — The control video is a neutral video with no content addressing back beliefs (fragility and need for protection).
  Arms: Control Video Education

SUMMARY:
In the current study we aim to evaluate the effects of a short educational video on improving the belief that "the back is fragile and needs to be protected" among the German speaking Swiss general population. We hypothesize that a short video education program can positively change the assessed back belief among the German speaking general population of Switzerland.

To evaluate the outcomes, we will use the 10-item version of the Back Pain Attitude Questionnaire (Back-PAQ). The primary outcome is the second question of the Back-PAQ-10 ("You could injure your back if you are not careful"). The secondary outcome of this study is the total score of the Back-PAQ-10.

The design of the present study is a two-group randomized controlled trial, with one intervention and one control group in a 1:1 allocation.

DETAILED DESCRIPTION:
This study will be conducted in collaboration with HESAV (Haute Ecole de Sante Vaud). The research group at the HESAV has developed an educational website in 2020, called "www.infomaldedos.ch". The website aims to educate people on low back pain, and common unhelpful beliefs about the back - primarily targeting the belief about the fragility of the back and the need for its protection - are addressed. In the current study we are going to translate the above-mentioned website to the German language. Furthermore, we are going to assess the quality and applicability of a short video intervention among the general population, using one of the videos from the website.

Participants will be recruited through social media and emails. A link will be created to the questionnaire and the educational video with LimeSurvey. A 'randomizer' built-in function will be used to blindly split people into intervention or control group. The link will be spread on social media platforms and through email. To induce a snowball sampling method, all participants will be asked to send the link further.

The length of the video intervention is 3 minutes. In the video, health care professionals, such as a psychologist, a medical doctor, a professor, and physiotherapist interviewed by a scientist explains the burden of LBP, how unhelpful beliefs affect treatment outcome, difficulties in the management of LBP and the optimal way of treating LBP. The scientist then inquires a representative patient about their own experiences of the management of LBP. At the end of the video the scientist encourages people to exercise despite LBP by performing various movements.

The control group will receive a neutral video about the back, selected from YouTube.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years

Exclusion Criteria:

* Professionals and students with prior knowledge on the topic of interest such as physiotherapists, osteopaths, and chiropractors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Sentiments about back vulnerability | One minute
  The primary outcome is the second question of the Back-PAQ-10 ("You could injure your back if you are not careful")

SECONDARY OUTCOMES:
Total Back-PAQ-10 score | Three minutes
  The secondary outcome of this study is the total score of the German version of the Back-PAQ-10.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schmid, PhD, Principal Investigator — Bern UAS
Locations (1):
- Bern University of Applied Sciences, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No